CLINICAL TRIAL: NCT04900662
Title: Patient Satisfaction and Visual Function Following Implantation of Trifocals or Extended
Brief Title: Patient Satisfaction and Visual Function Following Implantation of Trifocals or Extended Range of Vision Intraocular Lenses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Dr. Sherif R El-Defrawy, Clinician Scientist, University of Toronto
Other Study IDs: KEI20190718
Record Dates: First submitted 2020-10-06; First posted 2021-05-25 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Cataract
Keywords: cataract surgery; quality of life; preoperative fasting
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cataract surgery is a fast evolving refractive procedure, which aims to restore vision. The majority of intraocular lens (IOL) implants following cataract surgery are monofocal IOLs, which have been designed to improve distance vision by replacing the lens diopter power with a single focal point. Monofocal IOLs have been associated with very few complications related to the material or the technology. However, after the surgery patients are spectacle dependent for near and intermediate tasks. This, in turn, has decreased the patient's post-operative satisfaction and quality of life. Multifocal intraocular lenses (IOLs) were introduced into the market in the 1980s. This type of IOLs provides clear distance and near vision, which affects the quality of life and visual expectations of the patients who receive them. Studies have indicated higher levels of patient's satisfaction with regards to distance and near vision after the implantation of multifocal lenses. With Multifocal IOLs; however, patients are still spectacle dependent for intermediate tasks such as computer work. The recent development of trifocal IOLs has been found to provide optimal near, intermediate, and distance visual performances; decrease spectacle dependence; and increase patient satisfaction.AcrySof®IQ PanOptix™ (PanOptix) was introduced into the market in 2015 with a design that allows the IOL to provide optimal near, intermediate, and distance visual performances; decrease spectacle dependence; and increase patient satisfaction. Despite the benefits of corrected visual acuity at multiple distances, multifocal and/or trifocal IOLs are associated with certain disadvantages, including contrast sensitivity loss, dysphotopsia, halos and glare, which account for over a third of the justifications used for IOL model replacement. Dysphotopsia is the result of light reflecting off the intraocular lens (IOL) onto the retina which causes a variety of visual symptoms that are expressed in a positive or a negative form. Positive dysphotopsia refers to bright artifacts that are noticed in only certain lighting conditions, such as glare and halos. Negative dysphotopsia refers to the formation of a barrier, which prevents light from reaching the retina. The result of the negative form of dysphotopsia is the formation of shadows that are often in the temporal visual field. In 2014, the extended range of vision TECNIS Symfony®IOL (Symfony), with new optical technology using a proprietary achromatic diffractive echelette design, received a CE Mark. However, it was not until 2016 that this IOL became the first extended depth of focus (EDF) IOL to gain approval by the U.S. Food and Drug Administration. This new optical technology corrects the corneal chromatic aberration for enhanced contrast sensitivity, generating a continuous vision for distance through intermediate into near with low incidence of halos and glare. Despite the benefits of EDF IOLs, Monaco et al. conducted a study in Italy and indicated that both PanOptix and Symfony IOLs seemed to be good options for patients with intermediate-vision requirements, whereas the PanOptix IOL may be better for patients with near-vision requirements. A few studies in the literature have evaluated the performance of the PanOptix and Symfony IOLs in Europe. Our current study would add great value to the literature since to the best of our knowledge; this is the first study to address the same IOLs in North America. Cataract surgery expectations are continuously rising, and in an effort to maximize patient satisfaction post-operatively, the appropriateness of a patient for a particular IOL implantation should be evaluated carefully during the pre-operative assessment. Therefore, further research is warranted to evaluate patient satisfaction with both PanOptix and Symfony IOLs. The purpose of this study is to compare the visual outcomes and the subjective satisfaction results between patients implanted with PanOptix and Symfony IOLs.

ELIGIBILITY:
Inclusion Criteria:

- any patient receiving cataract surgery at KEI who is able and willing to participate over 18 years old.

Exclusion Criteria:

- less than 18, not receiving cataract surgery at KEI, not able or willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is patients receiving cataract surgery at KEI. Sampling is consecutive. No limitation based on gender or sex.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
patient burden from preoperative fasting | 2019-2021
  A questionnaire will be used to assess.
incidence of aspiration or cancellation of surgery because of preoperative fasting violation | 2019-2021
  A questionnaire will be used to assess.

CONTACTS AND LOCATIONS:
Locations (1):
- Kensington Eye Institute, Toronto, Ontario, Canada

REFERENCES:
- [Background] Calladine D, Evans JR, Shah S, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD003169. doi: 10.1002/14651858.CD003169.pub3. PMID 22972061
- [Background] de Medeiros AL, de Araujo Rolim AG, Motta AFP, Ventura BV, Vilar C, Chaves MAPD, Carricondo PC, Hida WT. Comparison of visual outcomes after bilateral implantation of a diffractive trifocal intraocular lens and blended implantation of an extended depth of focus intraocular lens with a diffractive bifocal intraocular lens. Clin Ophthalmol. 2017 Oct 26;11:1911-1916. doi: 10.2147/OPTH.S145945. eCollection 2017. PMID 29138533
- [Background] Santos BWL, Cançado JEP, Ferraz VAdS, Campos M. Evaluation of life quality of patients submitted to cataract surgery with implants of monofocal, bifocal and multifocal lenses. Revista Brasileira de Oftalmologia 2014;73:86-92
- [Background] Gundersen KG, Potvin R. Comparative visual performance with monofocal and multifocal intraocular lenses. Clin Ophthalmol. 2013;7:1979-85. doi: 10.2147/OPTH.S52922. Epub 2013 Oct 7. PMID 24143064
- [Background] Cochener B, Vryghem J, Rozot P, Lesieur G, Chevalier JP, Henry JM, David T, Lesueur L, Gatinel D, Ganem C, Blanckaert J, Van Acker E, Heireman S, Ghekiere S. Clinical outcomes with a trifocal intraocular lens: a multicenter study. J Refract Surg. 2014 Nov;30(11):762-8. doi: 10.3928/1081597X-20141021-08. PMID 25375849
- [Background] Attia MS, Auffarth GU, Khoramnia R, Linz K, Kretz FT. Near and intermediate reading performance of a diffractive trifocal intraocular lens using a reading desk. J Cataract Refract Surg. 2015 Dec;41(12):2707-14. doi: 10.1016/j.jcrs.2015.06.038. PMID 26796451
- [Background] Weeber HA, Meijer ST, Piers PA. Extending the range of vision using diffractive intraocular lens technology. J Cataract Refract Surg. 2015 Dec;41(12):2746-54. doi: 10.1016/j.jcrs.2015.07.034. PMID 26796456
- [Background] Escandon-Garcia S, Ribeiro FJ, McAlinden C, Queiros A, Gonzalez-Meijome JM. Through-Focus Vision Performance and Light Disturbances of 3 New Intraocular Lenses for Presbyopia Correction. J Ophthalmol. 2018 Jan 31;2018:6165493. doi: 10.1155/2018/6165493. eCollection 2018. PMID 29651343
- [Background] AcrySof [product information]. Fort Worth TAL, Inc.; 2015
- [Background] de Vries NE, Webers CA, Montes-Mico R, Tahzib NG, Cheng YY, de Brabander J, Hendrikse F, Nuijts RM. Long-term follow-up of a multifocal apodized diffractive intraocular lens after cataract surgery. J Cataract Refract Surg. 2008 Sep;34(9):1476-82. doi: 10.1016/j.jcrs.2008.05.030. PMID 18721706
- [Background] Kinard K, Jarstad A, Olson RJ. Correlation of visual quality with satisfaction and function in a normal cohort of pseudophakic patients. J Cataract Refract Surg. 2013 Apr;39(4):590-7. doi: 10.1016/j.jcrs.2012.11.023. Epub 2013 Feb 6. PMID 23395326
- [Background] Monaco G, Gari M, Di Censo F, Poscia A, Ruggi G, Scialdone A. Visual performance after bilateral implantation of 2 new presbyopia-correcting intraocular lenses: Trifocal versus extended range of vision. J Cataract Refract Surg. 2017 Jun;43(6):737-747. doi: 10.1016/j.jcrs.2017.03.037. PMID 28732606
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205